CLINICAL TRIAL: NCT06739902
Title: Comparing the Effectiveness of Traditional Physiotherapy Combined With Virtual Reality for Post-Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/770
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Traditional Physiotherapy Group
- Interventional group II (Active Comparator)
  Interventions: Combination Product: VR + Traditional Physiotherapy Group

INTERVENTIONS:
Diagnostic Test: Traditional Physiotherapy Group — Participants receive standard physiotherapy exercises aimed at improving motor function, balance, and trunk stability. These exercises include stretching, balance training, and muscle-strengthening activities.
  Arms: Interventional group I
Combination Product: VR + Traditional Physiotherapy Group — Participants receive the same physiotherapy exercises as the traditional group, but with additional sessions involving virtual reality exercises. The VR component includes immersive activities that stimulate motor control, coordination, and cognitive engagement to support functional recovery.
  Arms: Interventional group II

SUMMARY:
This study aims to evaluate the effectiveness of combining virtual reality (VR) therapy with traditional physiotherapy in post-stroke rehabilitation. Post-stroke patients often suffer from impairments in motor function, balance, and overall quality of life. While traditional physiotherapy is a widely accepted method for stroke recovery, incorporating VR technology may enhance treatment outcomes by providing an engaging, immersive environment that motivates patients to perform therapeutic movements.

DETAILED DESCRIPTION:
This study will compare the functional and quality-of-life improvements in patients undergoing traditional physiotherapy alone versus those receiving a combination of conventional physiotherapy and VR interventions. By assessing changes in motor function, trunk stability, balance, and quality of life, this research will provide valuable insights into whether VR can be an effective adjunctive tool in post-stroke rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Stroke, either ischemic or hemorrhagic
* Participants who can ambulate independently or with minimal assistance.
* Participants who were willing & able to adhere to the study protocol.
* Including participants who were attending follow-up appointments & completing outcome measures.
* Participants who were able to understand & provide written informed consent

Exclusion Criteria:

* Existence of additional neurological disorders (such as multiple sclerosis or Parkinson's disease) or serious medical conditions that could prevent participants from participating in the study.
* Participants receiving rehabilitation or rigorous physical treatment in the previous three months were excluded.
* Pregnant women or breastfeeding women.
* Participants who refused to participate in the study or provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 12 Months
  Assesses balance and stability.- *Purpose*: Assesses balance in older adults and individuals with balance disorders.
  * *Items*: 14 tasks, such as sitting, standing, reaching, and turning.
  * *Scoring*: Each task is scored on a scale of 0-4 (0 = inability to perform the task, 4 = normal performance).
  * *Total Score*: The maximum score is 56. Higher scores indicate better balance. A score below 45 indicates a higher risk of falling.
Trunk Impairment Scale (TIS) | 12 Months
  Measures trunk control and stability. SF-12 Health Survey: Evaluates quality of life in physical and mental health domains.The *Trunk Impairment Scale (TIS)* is a clinical tool used to assess trunk performance in individuals, particularly those with neurological impairments like stroke. It measures three key aspects: *static sitting balance, **dynamic sitting balance, and **coordination of trunk movements. The scale consists of **17 items*, with scores ranging from 0 to 23. Higher scores indicate better trunk control and stability. It helps clinicians evaluate and track improvements in trunk function over time, guiding rehabilitation interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital, Shadman 1, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No